CLINICAL TRIAL: NCT02304172
Title: The Efficacy and Safety of Thunderbeat in Thyroid Surgery: a Prospective Randomized Study
Brief Title: The Efficacy and Safety of Thunderbeat in Thyroid Surgery
Acronym: Thunderbeat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Olympus Korea Co., Ltd. (Unknown)
Responsible Party: Principal Investigator, Su-jin Kim, Clinical Assistant Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SNUHthyroid
Record Dates: First submitted 2014-11-20; First posted 2014-12-01 (Estimated); Last update posted 2016-02-15 (Estimated); Status verified 2016-02

CONDITIONS: Thyroid
Keywords: Thyroidectomy; Thunderbeat
MeSH Terms: conditions — Thyroid Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Thunderbeat (Group A) (Active Comparator): Patients submitted to thyroidectomy with the use of the Thunderbeat device.
  Interventions: Device: Thunderbeat (Group A)
- Harmonic (Group B) (Active Comparator): Patients submitted to thyroidectomy with the use of the Harmonic scalpel device
  Interventions: Device: Harmonic (Group B)

INTERVENTIONS:
Device: Thunderbeat (Group A) — hemostatic device utilized intraoperatively
  Arms: Thunderbeat (Group A)
Device: Harmonic (Group B) — hemostatic device utilized intraoperatively
  Arms: Harmonic (Group B)

SUMMARY:
The aim of this study is to compare the results of total thyroidectomy using the Thunderbeat device to that with the harmonic scalpel.

DETAILED DESCRIPTION:
Thunderbeat instrument combines an advanced bipolar clamp to the existing ultrasonic cutter. In the animal study with pig, the result of Thunderbeat shows fast abalation rate and same thermal conductivity. There has been reported a significant reduction in operative time and same complications with Thunderbeat in gynecology patient who underwent laparoscopic hysterectomy with lymph node dissection. Comparison of the utilization of this new device, however, with the Harmonic scalpel in thyroidectomy has not been performed in any study. The objective of this study is to compare the results of thyroidectomy using the Thunderbeat to that with the Harmonic scalpel device in respect to hemostasis, operative time and perioperative complications. All patients undergoing a thyroidectomy in our endocrine surgery department are randomized into those operated with Thunderbeat (Group A) and those with Harmonic scalpel (Group B).

ELIGIBILITY:
Inclusion Criteria:

* thyroidectomy
* normal vocal cord

Exclusion Criteria:

* additional surgical procedures together with the total thyroidectomy (i.e., parathyroidectomy or cervical lymph node dissection)
* Thyroid cancer patients with lymph node metastasis
* pregnant women
* uncontrolled hypertension, DM, chronic kidney failure, coagulation disorders
* aspirin or anti-platelet agent in 7 days
* Graves' disease or Hashimoto thyroiditis
* history of radiation treatment in head and neck area

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-11; Primary Completion 2015-12 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Postoperative complications including laryngeal nerve palsy, hypocalcemia, hemorrhage, hematoma, wound infection and skin burn | postoperatively (from the day of surgery until 3 months postoperatively)

SECONDARY OUTCOMES:
Hemostasis | intraoperatively (from skin incision to skin closure) & postoperatively (from skin closure until 2 day postoperatively)
Operative time | from skin incision to skin closure

CONTACTS AND LOCATIONS:
Overall Officials: Su-jin Kim, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided